CLINICAL TRIAL: NCT04081935
Title: Distraction Using Virtual Reality for Children During Intravenous Injections in an Emergency Department: A Randomized Trial
Brief Title: Distraction Using VR for Children During IV in an Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017B002
Record Dates: First submitted 2019-09-01; First posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2017-11

CONDITIONS: Pain; Fear
Keywords: school-age children, emergency treatment, intravenous placement, virtual reality, pain, fear
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduce pain and fair (Experimental): To determine whether the virtual reality as a distracting intervention could reduce pain and fear in school-age children receiving intravenous injections at an emergency department.
  Interventions: Device: Virtual Reality
- Compared (No Intervention): Normal treatment

INTERVENTIONS:
Device: Virtual Reality — virtual reality (VR) as a distracting intervention could reduce pain and fear during an IV placement for school-age children in the emergent department.
  Arms: Reduce pain and fair

SUMMARY:
Exploring the use of virtual reality as a distracting intervention strategy for school-age children to receive intravenous placement in emergency department, and further understand the effectiveness of reducing pain and fear during the invasive procedure.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 7-12
* Children who were clearly conscious
* Children who agreed and were required to receive intravenous injections after physicians' diagnoses
* Children and their primary caregivers who could communicate in Mandarin or Taiwanese
* Children and their primary caregivers who could read Chinese that agreed to participate in this study and sign written consent forms

Exclusion Criteria:

* Children with developmental delay, epilepsy, or heart diseases
* Children undergoing chemotherapy; children who were visually or hearing impaired
* Children who were nearsighted with more than 8.0 diopters or farsighted with 5.0 diopters
* Children who had sustained head trauma in the past month
* Children who were confirmed to be obese according to the recommended body mass index values for children and adolescents
* Children who required blood transfusions and blood preparation to be performed according to physician diagnoses
* Children who received two or more intravenous injections and had their blood drawn only one time

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
The degrees of pain experienced by the children. | The posttests 8 min after the tourniquets were worn.
  Measurement of pain using the Wong-Baker FACES Pain Rating Scale(WBFPS). The scale contains six cartoon faces showing pain ratings of 0-10, which are, from left to right, no pain (0), a little pain (2), mild pain (4), average pain (6), severe pain (8), and excruciating pain (10).The children, primary caregivers, and nurses were asked to select the faces that best described the pain levels experienced by the children receiving intravenous injections; the pain levels were subsequently converted into numerical values .
The degrees of fear experienced by the children. | The posttests 8 min after the tourniquets were worn.
  Measurement of fear using the Choldren Fear Scale(CFS).The scale consists of five cartoon faces showing fear ratings of 0-4, which were no fear (0), a little fear (1), some fear (2), very fear(3) and extreme fear (4). The children, primary caregivers, and nurses were asked to select the faces that best described the fear levels of the children receiving intravenous injections. The pain levels were subsequently converted into numerical values.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang-Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen YJ, Cheng SF, Lee PC, Lai CH, Hou IC, Chen CW. Distraction using virtual reality for children during intravenous injections in an emergency department: A randomised trial. J Clin Nurs. 2020 Feb;29(3-4):503-510. doi: 10.1111/jocn.15088. Epub 2019 Dec 4. PMID 31715039